CLINICAL TRIAL: NCT00005800
Title: A Phase II Neoadjuvant Trial of Sequential Doxorubicin and Docetaxel for the Treatment of Stage III Breast Cancer Measuring STAT Activation as a Predictor of Response to Therapy
Brief Title: Doxorubicin and Docetaxel in Treating Women With Stage III Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Aventis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-11971; CA 82533 (Other: NCI)
Record Dates: First submitted 2000-06-02; First posted 2003-10-08 (Estimated); Last update posted 2012-09-25 (Estimated); Status verified 2012-09

CONDITIONS: Breast Cancer
Keywords: stage IIIA breast cancer; stage IIIB breast cancer; inflammatory breast cancer
MeSH Terms: conditions — Breast Neoplasms; Inflammatory Breast Neoplasms | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; Docetaxel; Doxorubicin; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dose-Dense Chemotherapy (Experimental): Patients receive doxorubicin IV on day 1 every 2 weeks for 3 courses. After 3 weeks of rest, patients receive docetaxel IV over 1 hour on day 1 every 2 weeks for 3 courses. Filgrastim (G-CSF) is administered subcutaneously on days 3-10 of each doxorubicin and docetaxel course. Within 6 weeks of completion of neoadjuvant chemotherapy, patients undergo surgery with mastectomy or lumpectomy and axillary lymph node dissection.
  Interventions: Biological: Filgrastim; Drug: Docetaxel; Drug: Doxorubicin; Procedure: Surgery

INTERVENTIONS:
Biological: Filgrastim
  Other Names: G-CSF
Drug: Docetaxel
  Other Names: Taxotere®
Drug: Doxorubicin
  Other Names: doxorubicin hydrochloride; Adriamycin; Rubex
Procedure: Surgery — Within 6 weeks of completion of neoadjuvant chemotherapy, patients undergo surgery with mastectomy or lumpectomy and axillary lymph node dissection.

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of doxorubicin and docetaxel in treating women who have stage III breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the clinical and pathological response rate of sequential doxorubicin and docetaxel chemotherapy in the neoadjuvant treatment of women with stage III breast cancer.
* Measure signal transducer and activator of transcription (STAT) activation before and after this neoadjuvant chemotherapy regimen in this patient population.
* Correlate response to chemotherapy with STAT activation before and after this neoadjuvant chemotherapy regimen in these patients.
* Determine how other potential predictors of response correlate with STAT activation by measuring Bcl-2, Bcl-xL, Bax protein levels, tyrosine kinase levels, growth rate of the tumor, and apoptotic index before and after this neoadjuvant chemotherapy regimen in these patients.
* Correlate response to chemotherapy with levels of STAT activation in association with the presence of Bcl-2 proteins and tyrosine kinases, growth rate of the tumor, and apoptotic index in these patients.
* Evaluate the toxicity of this neoadjuvant chemotherapy regimen given in a dose-dense fashion in these patients.

OUTLINE: Patients receive doxorubicin IV on day 1 every 2 weeks for 3 courses. After 3 weeks of rest, patients receive docetaxel IV over 1 hour on day 1 every 2 weeks for 3 courses. Filgrastim (G-CSF) is administered subcutaneously on days 3-10 of each doxorubicin and docetaxel course. Within 6 weeks of completion of neoadjuvant chemotherapy, patients undergo surgery with mastectomy or lumpectomy and axillary lymph node dissection.

PROJECTED ACCRUAL: A total of 45 patients will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or pathologically confirmed stage III breast cancer

  * Clinical evidence of primary invasive breast tumor greater than 5 cm in dimension (T3) and no evidence of metastatic disease clinically or by staging studies including computed tomography (CT) scan of the chest, abdomen, and pelvis, and a bone scan
* Inflammatory breast carcinoma defined as diffuse brawny induration of the skin of the breast with an erysipeloid edge due to embolization of the dermal lymphatics and pathologic evidence of dermal lymphatic invasion
* No bilateral breast cancer unless synchronous
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 to 70

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* Eastern Cooperative Oncology Group (ECOG) 0-1

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin less than 2.0 mg/dL
* SGOT/SGPT less than 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase no greater than 4 times ULN provided SGOT/SGPT no greater than ULN

Renal:

* Creatinine no greater than 1.5 mg/dL

Cardiovascular:

* If prior cardiac event or ischemia on electrocardiogram, must be cleared by cardiologist
* LVEF at least 50% by resting MUGA
* No severe cardiac dysfunction
* No prior or concurrent angina pectoris, congestive heart failure, or major ventricular arrhythmias
* No uncontrolled essential hypertension

Other:

* Not pregnant or nursing
* Fertile patients must use effective nonhormonal barrier contraception
* No other prior malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or intraductal or lobular carcinoma in situ of the breast
* No other serious medical or psychiatric illness that would preclude study consent or treatment
* No prior severe and intolerable reactions to filgrastim (G-CSF)

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy to the breast

Surgery:

* Not specified

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 1999-04; Primary Completion 2006-01 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Pathological Response Rate | 7 years
  Evaluate the pathological response rate of sequential doxorubicin and docetaxel chemotherapy in the neoadjuvant treatment of women with stage III breast cancer. Pathologic response is classified as either complete pathologic response or partial pathologic response based on the size of residual tumor after treatment (complete pathologic response if 0 cm, partial pathologic response if >0 cm).

CONTACTS AND LOCATIONS:
Overall Officials: Susan Minton, D.O., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States